CLINICAL TRIAL: NCT01447901
Title: Prospective, Non-interventional, Non-randomised, Open-label, Adult Study to Assess the Long Term Biological Therapeutic Response to Alipogene Tiparvovec in Lipoprotein Lipase Deficiency (LPLD) and Comparing Postprandial Chylomicron Metabolism Following a Radiolabeled Meal in LPLD Subjects Previously Treated With Alipogene Tiparvovec (Studies CT-AMT-011-01 or -02) to Untreated LPLD Subjects (Study PREPARATION-02) and to Healthy Volunteers
Brief Title: Duration of Effect of Alipogene Tiparvovec Treatment, Which Was Administered in Other Studies
Status: Terminated | Type: Observational
Why Stopped: Business reason
Sponsor: Amsterdam Molecular Therapeutics (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-AMT-011-04
Record Dates: First submitted 2011-09-28; First posted 2011-10-06 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Hyperlipoproteinemia Type I
Keywords: Hyperlipoproteinemia Type I
MeSH Terms: conditions — Hyperlipoproteinemia Type I

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, faeces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- previously treated LPLD Cohort: Subjects in Cohort 1 (previously treated LPLD Cohort) must have received AMT-011 during Studies CT-AMT-011-01 or -02
- untreated LPLD control Cohort: Subjects in Cohort 2 (untreated LPLD control Cohort)) may have completed study PREPARATION-02 or known patients with genetically confirmed LPLD
- normal healthy control Cohort: Volunteers in Cohort 3 (normal healthy control Cohort) must not have LPLD

SUMMARY:
LPL (Lipoprotein Lipase) is an enzyme which plays an important role in the elimination of triglycerides (fat) and the clearance of dietary fat particles known as chylomicrons (CM) in the blood. In patients who have an abnormal LPL gene, the enzyme does not work (total, hereditary LPL deficiency), which results in a large increase in the amount of triglycerides (fats) and chylomicrons in the blood. This increases the risk of inflammation in the pancreas and leads to long term negative effects for bloods vessels (atherosclerosis). Current medications and / or a strict and low fat diet do not sufficiently reduce the level of triglycerides in order to prevent these conditions. To solve this problem, the company, AMT is developing a gene therapy (AMT-011).

In normal healthy individuals, fat particles are rapidly cleared from the circulation following a standard meal. Within approximately 3 hours the highest levels of fat is reached and clearance is achieved within the subsequent 9 hours. In LPLD subjects, the clearance of fat is greatly reduced as a direct consequence of the lack of LPL. During this study, a standard meal with a tracer (3H-palmitate) is given. Since palmitate is incorporated in the dietary fat, this study enabled monitoring of appearance of newly formed dietary fat into- and clearance of these newly formed dietary fats from the circulation, over time.

The principal aim of the study is to verify if the gene therapy (AMT 011) is still effective in the treatment of this condition. Systemic appearance and clearance of new formed dietary fat particles after ingestion of the meal will be determined by measuring the level of tracer at different time points.

DETAILED DESCRIPTION:
Lipoprotein lipase deficiency (LPLD) is a rare autosomal recessive inherited disorder caused by loss-of-function mutations in the lipoprotein lipase (LPL) gene. It is the most common genetic cause of hyperchylomicronaemia, a condition which results in continuous and excessively high levels of plasma chylomicrons (CM) and severe hypertriglyceridaemia. Lipoprotein lipase normally mediates the hydrolysis of triglycerides (TG) in CMs and very low-density lipoproteins (VLDL) and thereby aids in the clearance of TG-rich lipoproteins and reduction of TGs in the circulation.

Alipogene tiparvovec (Glybera®) is in development for the therapy of LPLD. In summary, alipogene tiparvovec contains the human lipoprotein (LPL) gene variant LPLS447X in a non-replicating vector in solution administered in a one-time series of intramuscular injections in the arms/legs.The aim of alipogene tiparvovec (Glybera®) administration is to provide LPL activity and to stimulate CM metabolism in LPLD patients.

To test the activity of LPL in subjects previously treated with alipogene tiparvovec in this study LPLD subjects will be given a radiolabeled meal supplemented with a labeled tracer, 3H-palmitate. Since dietary palmitate is incorporated into CMs as they are formed in the enterocytes of the gut, this enables monitoring of the appearance and subsequent clearance of newly formed CMs from the circulation over time, the so-called "postprandial test". The radiolabeled meal will be provided in a liquid form similar to a milkshake. After ingestion of the radiolabeled meal, level of radiolabel in the CM fraction at different time points prior to and during the postprandial phase will be measured and thus determine the appearance and clearance of CMs within the circulation.

The principal aim of the study is to increase the understanding of how long alipogene tiparvovec may be effective in the treatment of LPLD. To understand this, 3 cohorts of subjects will be studied: 1) Subjects with LPLD who have previously been treated with alipogene tiparvovec; 2) Subjects with LPLD who have not been treated with alipogene tiparvovec; and 3) Subjects who do not have LPLD (healthy volunteers). The subject's general state of health will also be monitored during the clinical study, and the possible disadvantages associated with the postprandial test will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided signed informed consent.
2. Male or female aged 18 to 70 years, inclusive at the time of consent.
3. Females of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable effective form of birth control from screening through Day 21 visit.
4. Subjects in Cohort 1 (previously treated LPLD Cohort) must have received AMT-011 during Studies CT-AMT-011-01 or -02 as verified by site personnel.
5. Subjects in Cohort 2 (untreated LPLD control Cohort)) may have completed study PREPARATION-02 as verified by site personnel or known patients with genetically confirmed LPLD.
6. Volunteers in Cohort 3 (normal healthy control Cohort) must not have LPLD.
7. Subjects must be in good general physical health with, in the opinion of the investigator, no other clinically significant and relevant abnormalities of medical history, and no abnormalities at the physical examination and routine laboratory evaluation performed prior to the study.
8. Must be able to communicate fully and effectively with the study personnel.

Exclusion Criteria:

1. Female subjects who have a positive serum pregnancy test or who are nursing.
2. Known allergy to any of the constituents of the radiolabeled meal/radio labeled agent, or a history of severe allergic or anaphylactic reactions.
3. Investigator-determined clinically significant disease (other than LPLD for those subjects with LPLD), that would affect the subject's participation in the study.
4. Healthy Volunteers with a history or presence of neurological, haematological, psychiatric, gastrointestinal, pulmonary, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs, including plasma lipids out side normal range for age and gender and a body mass index (BMI) >30.
5. Any current or relevant previous history of serious, severe, or unstable physical or psychiatric illness, any medical disorder that may make the participant unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.
6. A laboratory value at screening outside the normal range unless it is judged by the investigator as not clinically significant after appropriate evaluation.
7. Clinically significant ECG at screening as determined by the investigator.
8. Blood donations (≥1 unit) during the 2 months preceding and following the study or other significant blood loss.
9. Other unspecified reasons that, in the opinion of the investigator or sponsor, make the subject unsuitable for enrolment.
10. Any individual involved in the planning or conduct of this study. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Lipoprotein Lipase Deficiency (LPLD) Patients
  * Healthy volunteers (community sample)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacodynamics | pre dose, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24 hours post dose
  Peak level, time-to-peak, and area under the curve (AUC) for tracer in plasma and chylomicron (CM) fraction to assess metabolism of newly-formed CMs in LPLD subjects previously treated with alipogene tiparvovec and to compare with untreated LPLD subjects and healthy controls.

SECONDARY OUTCOMES:
Triglyceride (TG)-rich lipoproteins | pre dose, 0, 1, 2, 3, 4, 4, 6, 7, 8, 9, 12, 24 hours post dose
  Surface and core components of TG-rich lipoproteins (TG, TChol, apoB100, and apoB48)in plasma and in the CM fraction will be measured.
Glucose | pre dose, 0, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24 hours post dose
  The levels of glucose in plasma.
Adverse Events (AE) | Up to 21 days. Serious AEs will be followed to their resolution.
  Monitoring general state of health of subjects and to assess the safety of ingestion of a radiolabeled meal, containing the radiolabel 3H palmitate through review of the incidence and severity of adverse events (AEs).
Laboratory tests | Up to 21 days
  Monitoring general state of health in LPLD subjects previously treated with alipogene tiparvovec compared to untreated LPLD subjects and healthy volunteers through review of laboratory findings (haematology, clinical chemistry, and urinalysis).
Vital signs | Up to 21 days
  To monitor the general state of health in LPLD subjects previously treated with alipogene tiparvovec compared to untreated LPLD subjects and healthy volunteers through review of the vital signs.
Physical examination | Up to 21 days
  To monitor the general state of health in LPLD subjects previously treated with alipogene tiparvovec compared to untreated LPLD subjects and healthy volunteers through review of physical examination findings.
ECG | Up to 21 days
  To monitor the general state of health in LPLD subjects previously treated with alipogene tiparvovec compared to untreated LPLD subjects and healthy volunteers through review of 12-lead electrocardiograms (ECGs).
C-peptide | pre dose, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24 post dose
  Levels of C-peptide in plasma
Non Esterified Fatty Acids (NEFA) | pre dose, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24 post dose
  Levels of NEFA in plasma will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gaudet, MD PhD, Principal Investigator — ECOGENE-21 Clinical Trial Center
Locations (1):
- ECOGENE-21 Clinical Trial Center, Chicoutimi, Quebec, Canada

REFERENCES:
- [Background] Bickerton AS, Roberts R, Fielding BA, Hodson L, Blaak EE, Wagenmakers AJ, Gilbert M, Karpe F, Frayn KN. Preferential uptake of dietary Fatty acids in adipose tissue and muscle in the postprandial period. Diabetes. 2007 Jan;56(1):168-76. doi: 10.2337/db06-0822. PMID 17192479
- [Background] Black DM, Sprecher DL. Dietary treatment and growth of hyperchylomicronemic children severely restricted in dietary fat. Am J Dis Child. 1993 Jan;147(1):60-2. doi: 10.1001/archpedi.1993.02160250062018. PMID 8418601
- [Background] Chait A, Brunzell JD. Chylomicronemia syndrome. Adv Intern Med. 1992;37:249-73. PMID 1557997
- [Background] Fortson MR, Freedman SN, Webster PD 3rd. Clinical assessment of hyperlipidemic pancreatitis. Am J Gastroenterol. 1995 Dec;90(12):2134-9. PMID 8540502
- [Background] Miles JM, Park YS, Walewicz D, Russell-Lopez C, Windsor S, Isley WL, Coppack SW, Harris WS. Systemic and forearm triglyceride metabolism: fate of lipoprotein lipase-generated glycerol and free fatty acids. Diabetes. 2004 Mar;53(3):521-7. doi: 10.2337/diabetes.53.3.521. PMID 14988233
- [Background] Normand-Lauziere F, Frisch F, Labbe SM, Bherer P, Gagnon R, Cunnane SC, Carpentier AC. Increased postprandial nonesterified fatty acid appearance and oxidation in type 2 diabetes is not fully established in offspring of diabetic subjects. PLoS One. 2010 Jun 4;5(6):e10956. doi: 10.1371/journal.pone.0010956. PMID 20532041
- [Background] Rip J, Nierman MC, Ross CJ, Jukema JW, Hayden MR, Kastelein JJ, Stroes ES, Kuivenhoven JA. Lipoprotein lipase S447X: a naturally occurring gain-of-function mutation. Arterioscler Thromb Vasc Biol. 2006 Jun;26(6):1236-45. doi: 10.1161/01.ATV.0000219283.10832.43. Epub 2006 Mar 30. PMID 16574898
- [Background] Rip J, Nierman MC, Sierts JA, Petersen W, Van den Oever K, Van Raalte D, Ross CJ, Hayden MR, Bakker AC, Dijkhuizen P, Hermens WT, Twisk J, Stroes E, Kastelein JJ, Kuivenhoven JA, Meulenberg JM. Gene therapy for lipoprotein lipase deficiency: working toward clinical application. Hum Gene Ther. 2005 Nov;16(11):1276-86. doi: 10.1089/hum.2005.16.1276. PMID 16259561
- [Background] Ross CJ, Twisk J, Bakker AC, Miao F, Verbart D, Rip J, Godbey T, Dijkhuizen P, Hermens WT, Kastelein JJ, Kuivenhoven JA, Meulenberg JM, Hayden MR. Correction of feline lipoprotein lipase deficiency with adeno-associated virus serotype 1-mediated gene transfer of the lipoprotein lipase S447X beneficial mutation. Hum Gene Ther. 2006 May;17(5):487-99. doi: 10.1089/hum.2006.17.487. PMID 16716106
- [Background] Santamarina-Fojo S. The familial chylomicronemia syndrome. Endocrinol Metab Clin North Am. 1998 Sep;27(3):551-67, viii. doi: 10.1016/s0889-8529(05)70025-6. PMID 9785052
- [Background] Wittrup HH, Tybjaerg-Hansen A, Nordestgaard BG. Lipoprotein lipase mutations, plasma lipids and lipoproteins, and risk of ischemic heart disease. A meta-analysis. Circulation. 1999 Jun 8;99(22):2901-7. doi: 10.1161/01.cir.99.22.2901. PMID 10359734
- See also: Homepage Sponsor — http://www.amtbiopharma.com/